CLINICAL TRIAL: NCT01158118
Title: A Phase II Trial Evaluating the Safety and Efficacy of Plerixafor and Sargramostim (GM-CSF) for the Mobilization of Peripheral Blood Stem Cells (PBSC) From Normal, HLA-Matched Allogeneic Sibling Donors
Brief Title: Plerixafor and Sargramostim (GM-CSF) for Mobilization of Allogeneic Sibling Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-1154 / 201108083
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma
Keywords: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Donor (Experimental): Days 1-5: Mobilization with 5 mcg/kg/day GM-CSF (first 4 donors were mobilized with 10 mcg/kg GM-CSF then changed to 5 mcg/kg for remaining donors)
  Day 5: Mobilization with 320 mcg/kg plerixafor IV
  Day 5: Leukopheresis
  If PBSC collected are not adequate, then donor will be mobilized with GM-CSF and plerixafor IV on day 6 and have leukopheresis collection on day 6.
  Interventions: Drug: Sargramostim; Drug: Plerixafor
- Arm 2 - Recipient (No Intervention): Conditioning Regimens
  * fludarabine and busulfan +/- thymoglobulin
  * fractionated total body irradiation and cyclophosphamide
  * busulfan and cyclophosphamide
  * single dose total body irradiation and cyclophosphamide
  Day -2 = GvHD prophylaxis
  Day 0 or +1 = PBSC transplant
  Day +7 until neutrophil engraftment = G-CSF 5 ug/kg/day

INTERVENTIONS:
Drug: Sargramostim
  Other Names: GM-CSF, Leukine
  Arms: Arm 1 - Donor
Drug: Plerixafor
  Other Names: AMD3100, Mozobil
  Arms: Arm 1 - Donor

SUMMARY:
This study will gather information about the combination the drugs plerixafor with sargramostim in donors of blood-forming cells (stem cells). These stem cells will be collected from the donor and transplanted into their sibling. The investigators believe that the two drugs together will provide enough stem cells for transplantation and may also reduce the risk of graft versus host disease.

DETAILED DESCRIPTION:
The main purpose of this study is to gather information about the combination the drugs plerixafor with sargramostim in donors of blood-forming cells (stem cells). Stem cells can be taken from the bone marrow of the pelvic bones or from the blood following treatment with drugs called growth factors; sargramostim is such a drug. Once stem cells leave the bone marrow and circulate in the blood, they are called peripheral blood stem cells (PBSCs). These cells can be collected through a routine procedure called apheresis, which involves placing two IVs into the arm which are connected to an apheresis machine; the machine then takes blood from the body, removes the stem cells, and returns the blood to the body.

Normally, a growth factor called filgrastim is given to donors in order to collect the stem cells used for transplantation. However, when stem cells collected using filgrastim are transplanted in patients, a possible unpredictable complication is graft versus host disease. It's thought that using a different growth factor such as sargramostim might reduce the occurrences of graft versus host disease in patients. However, sargramostim alone does not provide as many stem cells for transplantation as other growth factors. Plerixafor is another drug that can increase the number of PBSCs in a donor, but like with sargramostim, plerixafor alone does not always provide enough stem cells. This is why sargramostim and plerixafor are being combined in this study: the investigators believe that the two drugs together will provide enough stem cells for transplantation and may also reduce the risk of graft versus host disease.

ELIGIBILITY:
Inclusion Criteria:

Donor Eligibility

* Donor is 18 to 65 years of age inclusive.
* If female and of child-bearing age, donor must be non-pregnant, not breastfeeding, and agree to use adequate contraception.
* Donor is a 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* Donor has adequate cardiac function with no history of congestive heart failure and no history of atrial fibrillation or ventricular tachyarrhythmia.
* Donor has adequate renal function as defined by a calculated serum creatinine clearance of ≥56 ml/min for females and ≥64 ml/min for males.
* Donor has adequate hepatic function as defined by a total bilirubin <2x normal or absence of hepatic fibrosis/cirrhosis.
* Donor has adequate neurologic function as defined by NO evidence of a severe central or peripheral neurologic abnormality. No history of cerebrovascular accident or seizure disorder requiring anticonvulsant medication.
* Donor must be HIV-1&2 antibody and HTLV-I&II antibody sero-negative, by FDA licensed test.
* Donor must have an ECOG performance status of 0 or 1.
* Donor must demonstrate ability to be compliant with study regimen.
* Donor must not have an active infection at the time of study entry.
* Donor does not have active alcohol or substance abuse within 6 months of study entry.
* Donor is not currently enrolled on another investigational agent study.
* Donor does not have any medical condition, which, in the opinion of the clinical investigator, would interfere with his/her evaluation.
* Ability of the donor to understand and the willingness to sign a written informed consent document.

Recipient Eligibility

* Recipient must have available the successful collection of a GM-CSF + plerixafor mobilized product. When an adequate collection cannot be obtained, G-CSF will be used and some recipients may need to receive a combined product of mobilized cells with plerixafor + GM-CSF and G-CSF mobilized cells. Recipients who receive less than 2.0 X 106 CD34+ cells/kg/actual recipient weight after six days of GM-CSF and two days of IV plerixafor will not be considered "eligible" but followed per protocol for safety purposes only.
* Recipient is 18 to 65 years of age inclusive.
* Recipient is willing and has a 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* Recipient must provide signed informed consent.
* If female and of child-bearing age, recipient must be non-pregnant, not breastfeeding, and using adequate contraception.
* Recipient must have one of the following diagnoses:

  * Acute myelogenous leukemia (AML) in 1st or subsequent remission or in relapse,
  * Acute lymphoblastic leukemia (ALL) in 1st or subsequent remission or in relapse,
  * Myelodysplastic syndrome either intermediate 1 or 2, or high risk by the International Prognostic Scoring System,
  * Chronic myelogenous leukemia (CML) in accelerated or second chronic phase,
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete remission, partial remission, or refractory relapse,
  * Chronic lymphocytic leukemia (CLL), Rai Stage 2-4, failing at least 2 prior regimens, OR
  * Multiple myeloma (MM), Stage 2-3.
  * Myeloproliferative disorder or neoplasm
* Recipient must have adequate cardiac function with a left ventricular ejection fraction ≥ 40%.
* Recipient must have adequate pulmonary function defined as NO severe or symptomatic restrictive or obstructive lung disease, and formal pulmonary function testing showing an FEV1 ≥50% of predicted and a DLCO ≥40% of predicted, corrected for hemoglobin.
* Recipient must have adequate renal function as defined by a serum creatinine clearance (Cockcroft-Gault equation)of ≥56 ml/min for females and ≥64 ml/min for males of normal
* Recipient must have adequate hepatic function as defined by a total bilirubin <2x normal or absence of hepatic fibrosis/cirrhosis.
* Recipient must have adequate neurologic function as defined by NO evidence of a severe central or peripheral neurologic abnormality. Patients with a history of previous CNS tumor involvement are eligible provided they are without symptoms or signs and the CNS is now free of disease on lumbar puncture and CT scan of the brain.
* Recipient must have no evidence of active infection at the time of the transplant preparative regimen or at time of transplantation.
* Recipient must be HIV-1&2 antibody and HTLV-I & II antibody sero-negative, by FDA licensed test.
* Recipient has an ECOG performance status of 0 or 1.
* Recipient must demonstrate ability to be compliant with medical regimen.
* Recipient must not have active alcohol or substance abuse within 6 months of study entry.
* Recipient must not be enrolled on another investigational agent concurrently.
* Recipient must not have any medical condition, which, in the opinion of the clinical investigator, would interfere with the evaluation of the patient.
* Recipient must have a life expectancy of greater than 4 weeks.
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

Donor Exclusion Criteria in addition to that stated above

* Donor may not be receiving any other investigational agents.
* Donor may not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to plerixafor or GM-CSF, or known hypersensitivity to yeast-derived products or any component of the product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Started | 24 | 24
Completed | 23 | 21
Not Completed | 1 | 3
Not completed — Screen failure | 1 | 0
Not completed — Donor match was a screen failure | 0 | 1
Not completed — Suffered stroke prior to transplant | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Median (Full Range); unit: years] | 53 [21 to 65] | 57 [32 to 64] | 56 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 11 | 16 | 27
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Donors Requiring a Second Collection to Obtain a Minimum CD34/Kg (2 x 10^6) Necessary for Allogeneic Stem Cell Transplantation
Description: The primary endpoint is to reduce the number of donors treated with GM-CSF who require a second collection to obtain a minimum CD34/Kg (2 x 106) necessary for allogeneic stem cell transplantation when compared to historic controls mobilized with GM-CSF or plerixafor alone. A reduction in failed first leukapheresis from 40% to less than 10% as seen with G-CSF alone would be considered clinically meaningful.
Time Frame: Up to 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Donor
Number analyzed (Participants) | 23
Participants | 4

2. Secondary Outcome: Proportion of Donors Who Experience Grade 3-4 Infusion Toxicity
Description: Infusional toxicity will be evaluated by measuring the patient's blood pressure, heart rate, respirations and temperature one hour prior to the allograft infusion and then 15 minutes, 30 minutes, one hour, 2 hours, and 4 hours, and 6 hours post infusion. Donors will have vital signs collected at each time point. EKGs will be performed immediately prior to IV AMD3100 and one hour after infusion.
Time Frame: 30 days after completion of therapy (estimated to be 36 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Donor
Number analyzed (Participants) | 23
Participants | 2

3. Secondary Outcome: Number of Donors Who Mobilize ≥ 2x10^6 CD34+ Cells/Kg Recipient Weight Safely Following One or Two Aphereses
Description: -The donor will undergo a leukapheresis procedure to process 20L of blood volume. After the procedure, the collection will be analyzed to look at CD34+ cell content. If it contains at least 2x10^6 CD34+ cells/kg, then the procedure will be considered successful.
Time Frame: Up to 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Donor
Number analyzed (Participants) | 23
Participants | 23

4. Secondary Outcome: Percentage of Donors Who Reach 5x10^6 CD34+ Cells/Kg Recipient Weight in 1 or 2 Aphereses
Description: -The donor will undergo a leukapheresis procedure to process 20L of blood volume. After the procedure, the collection will be analyzed to look at CD34+ cell content. The percentage of donors who reach at least 5x10^6 CD34+ cells/Kg recipient weight will be analyzed for this outcome measure.
Time Frame: 6 days
Population: -If patients achieved ≥ 2x10^6 CD34+ cells/Kg, they were not required to go on to a second day of collection
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Donor
Number analyzed (Participants) | 23
Participants | 8

5. Secondary Outcome: Determine if Peripheral Blood Stem Cell Products Collected After Mobilization With IV Plerixafor Can be Used Safely for Hematopoietic Cell Transplantation in HLA-matched Recipients as Measured by Time to Neutrophil Engraftment (Recipient Only)
Description: -Time to neutrophil engraftment is measured by determining the first of 3 consecutive measurements of neutrophil count ≥ 500/ul following conditioning regimen induced nadir.
Time Frame: Up to Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 21
Participants | 20

6. Secondary Outcome: Kinetics of Immune Reconstitution as Measured by Time to Neutrophil Engraftment (Recipient Only)
Description: as for outcome 5
Time Frame: Up to Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 21
days | 12 [11 to 22]

7. Secondary Outcome: Kinetics of Immune Reconstitution as Measured by Time to Platelet Engraftment (Recipient Only)
Description: -Time to platelet engraftment is measured by determining the first of 3 consecutive measurements of platelet count ≥ 20,000/ul without platelet transfusion support for 7 days.
Time Frame: Up to Day 180
Population: 1 recipient did not have platelet engraftment by Day 180 and is not evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 20
days | 22 [15 to 106]

8. Secondary Outcome: Rate of Acute Graft vs. Host Disease (GvHD) (Recipient Only)
Description: -Incidence and severity of acute GVHD will be assessed based on the Seattle criteria. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Time Frame: Up through Day 100
Population: 3 of the recipients received cells mobilized by 10 mcg/kg of GM-CSF and the 11 recipients received stem cells from donors mobilized with the decreased dose of 5 mcg/kg of GM-CSF.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 21
Participants | 14

9. Secondary Outcome: Rate of Chronic Graft vs. Host Disease (GvHD) (Recipient Only)
Description: Incidence and severity of chronic GVHD will be assessed based on the NIH consensus criteria and global severity scoring system. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Time Frame: Day 100-1 year
Population: 6 participants are not evaluable for this outcome measure as they came off study prior to the start of chronic GvHD assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 15
Participants | 10

10. Secondary Outcome: Transplant Related Mortality (Recipient Only)
Description: Death that results from a transplant procedure related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 21
Participants | 2

11. Secondary Outcome: Relapse and Disease Progression Rate
Description: -A patient will be considered relapsed (disease progressed) when there is a recurrence of the original malignant disease after transplantation.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 21
Participants | 5

12. Secondary Outcome: Death of Any Cause (Recipients Only)
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2 - Recipient
Number analyzed (Participants) | 21
Participants | 9

ADVERSE EVENTS:
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Serious Adverse Events (participants affected / at risk) | 1/23 | 8/21
Other Adverse Events (participants affected / at risk) | 23/23 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Donor (N=23) | Arm 2 - Recipient (N=21)
Cardiac arrest (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rigors (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Transamintis (Investigations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Donor (N=23) | Arm 2 - Recipient (N=21)
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 6
Alkaline phosphatase increased (Investigations) | 0 | 3
Allergic reaction (Immune system disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 11 | 7
Anorexia (Metabolism and nutrition disorders) | 3 | 7
Anxiety (Psychiatric disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Bloating (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Catheter site swelling (General disorders) | 0 | 1
Catheter site tenderness (General disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Chills (General disorders) | 0 | 4
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Creatinine increased (Investigations) | 1 | 6
Depression (Psychiatric disorders) | 1 | 1
Diaphoresis (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 17
Dislocation Left Hip Hemiarthroplasty (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 9
Ejection fraction decreased (Investigations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Esophageal pain (Gastrointestinal disorders) | 0 | 1
Excessive dreams (Psychiatric disorders) | 0 | 1
Facial pain (General disorders) | 1 | 2
Fall (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (General disorders) | 9 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 9
Fever (General disorders) | 1 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flu-like symptoms (General disorders) | 3 | 0
Flushing (Vascular disorders) | 1 | 1
GVHD - Skin (Rash) (Skin and subcutaneous tissue disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Gum infection (Infections and infestations) | 0 | 1
HSV stomatitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 9 | 10
Heart failure (Cardiac disorders) | 0 | 1
Heart racing (Cardiac disorders) | 0 | 1
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 6
Hypernatremia (Investigations) | 0 | 2
Hypersomnia (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 5
Hyperuricemia (Investigations) | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 5
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Vascular disorders) | 5 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
INR increased (Investigations) | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Injection site reaction (General disorders) | 7 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Jaundice (Skin and subcutaneous tissue disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Left chest fasciculations (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 2
Lymphocyte count increased (Investigations) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Nail infection (Infections and infestations) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 8 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 8
Non-cardiac chest pain (General disorders) | 2 | 4
Oral HSV (Infections and infestations) | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Pain at catheter placement site (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Palpitations (Cardiac disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 4 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Phosphate increased (Metabolism and nutrition disorders) | 0 | 1
Platelet count decreased (Investigations) | 14 | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Presyncope (Nervous system disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash - GVHD (Chest) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash - GVHD (Palms) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash - GVHD (Skin in general) (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 7
Rectal pain (Gastrointestinal disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 3 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 2
Skin infection (Infections and infestations) | 1 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 3
Somnolence (Nervous system disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Stool VRE (Infections and infestations) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tonsilitis (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 7 | 0
Visual disturbance (purple lights) (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4
White blood cell count decreased (Investigations) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes